CLINICAL TRIAL: NCT01914120
Title: A Multicenter, Observational, Phase III Clinical Study: the Quality of Life Assessment of Lung Cancer Patients in China.
Brief Title: the Quality of Life Assessment of Lung Cancer Patients in China
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Li Zhang, Profressor, Sun Yat-sen University
Other Study IDs: QLQ-CN
Record Dates: First submitted 2013-07-28; First posted 2013-08-01 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Lung Cancer
Keywords: lung cancer; quality of life; FACT-L
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal of this study is assess the quality of life of advanced non-small cell lung cancer (NSCLC) patients who are undergoing first-line chemotherapy, analyze the current status and tendency of quality of life (QOL). The method is to use the Functional Assessment of Cancer Therapy-Lung (FACT-L) scales, assess the quality of life before the chemotherapy, after 1st cycle of chemotherapy and after 2nd cycle. After 3 time-points, investigators analyze all the subscales and constructs of FACT-L. The assumption is the quality of life will be better after 2 cycle of chemotherapy.

DETAILED DESCRIPTION:
1. Lung cancer is the most deadly cancer in the world, 85% lung cancer are non-small cell lung cancer (NSCLC). The quality of life of NSCLC patients become more and more important, because of most NSCLC is incurable.
2. The recruitment will take place in 20 center all over the country and 500 patients will enrolled.

ELIGIBILITY:
Inclusion Criteria:

* age: >18 and <75 years old
* pathological or cytological diagnosis confirmed advanced non-small cell lung cancer
* Eastern Cooperative Oncology Group Performance Status: 0-2
* have never receive any kind of anti-cancer chemotherapy
* agree to regularly assessment of quality of life
* sign the informed consent form

Exclusion Criteria:

* Currently attending any antitumor drug clinical trials
* Pregnancy or breast-feeding women
* Currently receiving anti-tumor chemotherapy, or received any antitumor chemotherapy previously.
* not suitable to participate in this test

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced non-small cell lung cancer patients diagnosed by pathological or cytological methods, and also have a imageological diagnosis within 6 weeks for clinical staging.
  Clinical stage IIIB or IV. Chemo-naive patients: have never receive any kind of anti-cancer chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2012-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
the change of quality of life | Change from baseline quality of life at 6 weeks
  use Functional Assessment of Cancer Therapy-Lung (FACT-L) scales assess the quality of life to all subjects.
  before chemotherapy; after 1st chemotherapy; after 2nd chemotherapy;

SECONDARY OUTCOMES:
overall survival | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Professor, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Shi Y, Xing P, Fan Y, Zhang X, Hu C, Wang C, Liu X, Chen X, Zhou J, Wang M, Wu M, Han B, Fan M. Current small cell lung cancer treatment in China. Thorac Cancer. 2015 May;6(3):233-8. doi: 10.1111/1759-7714.12218. Epub 2015 Jan 15. PMID 26273367
- [Background] Zell JA, Ignatius Ou SH, Ziogas A, Anton-Culver H. Validation of the proposed International Association for the Study of Lung Cancer non-small cell lung cancer staging system revisions for advanced bronchioloalveolar carcinoma using data from the California Cancer Registry. J Thorac Oncol. 2007 Dec;2(12):1078-85. doi: 10.1097/JTO.0b013e31815ba260. PMID 18090578
- [Background] Hopwood P, Stephens RJ. Symptoms at presentation for treatment in patients with lung cancer: implications for the evaluation of palliative treatment. The Medical Research Council (MRC) Lung Cancer Working Party. Br J Cancer. 1995 Mar;71(3):633-6. doi: 10.1038/bjc.1995.124. PMID 7533520
- [Background] Lutz S, Norrell R, Bertucio C, Kachnic L, Johnson C, Arthur D, Schwarz M, Palardy G. Symptom frequency and severity in patients with metastatic or locally recurrent lung cancer: a prospective study using the Lung Cancer Symptom Scale in a community hospital. J Palliat Med. 2001 Summer;4(2):157-65. doi: 10.1089/109662101750290191. PMID 11441624
- [Background] Vainio A, Auvinen A. Prevalence of symptoms among patients with advanced cancer: an international collaborative study. Symptom Prevalence Group. J Pain Symptom Manage. 1996 Jul;12(1):3-10. doi: 10.1016/0885-3924(96)00042-5. PMID 8718910
- [Background] Temel JS, Greer JA, Muzikansky A, Gallagher ER, Admane S, Jackson VA, Dahlin CM, Blinderman CD, Jacobsen J, Pirl WF, Billings JA, Lynch TJ. Early palliative care for patients with metastatic non-small-cell lung cancer. N Engl J Med. 2010 Aug 19;363(8):733-42. doi: 10.1056/NEJMoa1000678. PMID 20818875
- [Background] Splinter TA. Chemotherapy in advanced non-small cell lung cancer. Eur J Cancer. 1990;26(10):1093-9. doi: 10.1016/0277-5379(90)90059-3. PMID 2177347
- [Background] Cella DF, Bonomi AE, Lloyd SR, Tulsky DS, Kaplan E, Bonomi P. Reliability and validity of the Functional Assessment of Cancer Therapy-Lung (FACT-L) quality of life instrument. Lung Cancer. 1995 Jun;12(3):199-220. doi: 10.1016/0169-5002(95)00450-f. PMID 7655830
- [Background] Hollen PJ, Gralla RJ, Kris MG, Cox C. Quality of life during clinical trials: conceptual model for the Lung Cancer Symptom Scale (LCSS). Support Care Cancer. 1994 Jul;2(4):213-22. doi: 10.1007/BF00365725. PMID 8087439
- [Background] Cella D, Eton DT, Fairclough DL, Bonomi P, Heyes AE, Silberman C, Wolf MK, Johnson DH. What is a clinically meaningful change on the Functional Assessment of Cancer Therapy-Lung (FACT-L) Questionnaire? Results from Eastern Cooperative Oncology Group (ECOG) Study 5592. J Clin Epidemiol. 2002 Mar;55(3):285-95. doi: 10.1016/s0895-4356(01)00477-2. PMID 11864800
- [Derived] Liu J, Ma Y, Gao R, Liu X, Wang Y, Yu J, Zhan J, Huang Y, Qin H, Zhang L. Prognostic effects of health-related quality of life at baseline and early change in health-related quality of life on response to treatment and survival in patients with advanced lung cancer: a prospective observational study in China. BMJ Open. 2022 Feb 14;12(2):e047611. doi: 10.1136/bmjopen-2020-047611. PMID 35165103